CLINICAL TRIAL: NCT07384195
Title: A Phase III Study to Assess Efficacy and Safety of N-Acetyl-GED-0507-34-LEVO Gel 5%, Applied Once Daily for 12 Weeks in Patients With Acne Vulgaris (GEDACNE-1)
Brief Title: A Study to Assess Efficacy and Safety of N-Acetyl-GED-0507-34-LEVO Gel 5%, in Patients With Acne Vulgaris (GEDACNE-1)
Acronym: GEDACNE-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: PPM Services S.A. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAC-GED-0507-ACN-01-23-A; 2023-510339-12-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-12; First posted 2026-02-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-10

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N-Acetyl-GED-0507-34-Levo 5% gel (Experimental)
  Interventions: Drug: N-Acetyl-GED-0507-34-Levo 5% gel
- N-Acetyl-GED-0507-34-Levo corresponding vehicle (Placebo Comparator)
  Interventions: Drug: N-Acetyl-GED-0507-34-Levo corresponding vehicle

INTERVENTIONS:
Drug: N-Acetyl-GED-0507-34-Levo 5% gel — Each patient will apply a fingertip unit of N-Acetyl-GED-0507-34-Levo 5% gel as a thin film, once daily (OD), to the entire facial skin area and the affected skin areas of the trunk accessible for self-application (i.e., shoulders, upper back, and upper anterior chest) for 12 consecutive weeks.
  Arms: N-Acetyl-GED-0507-34-Levo 5% gel
Drug: N-Acetyl-GED-0507-34-Levo corresponding vehicle — Each patient will apply a fingertip unit of N-Acetyl-GED-0507-34-Levo corresponding vehicle as a thin film, once daily (OD), to the entire facial skin area and the affected skin areas of the trunk accessible for self-application (i.e., shoulders, upper back, and upper anterior chest) for 12 consecutive weeks.
  Other Names: Placebo
  Arms: N-Acetyl-GED-0507-34-Levo corresponding vehicle

SUMMARY:
The clinical trial aims to test a new drug for acne vulgaris. The trial is performed to answer this question "Is it possible to reduce the number of skin lesions on your face/trunk, after daily applications for 12 consecutive weeks of a new drug?". The trial aims to accurately measure the effects of the new treatment (N-Acetyl-GED-0507-34-LEVO gel 5%) and to achieve this, patients will be randomly assigned to one of the following treatments:

* Study drug 1: test item, containing active ingredient
* Study drug 2: a preparation not containing any active ingredient (vehicle). Researchers will compare active to vehicle to see if there are differences in the efficacy.

Participants will:

* Apply drug or a placebo every day for 12 weeks
* Visit the site once every 4 weeks for checkups and tests (where applicable)
* Record on a diary the daily applications of the study drug at home, and record any adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained: Written informed consent, before any study-related procedure, personally signed and dated by the patient if the patient is ≥ 18 years old, or signed and dated by the parents or the legal guardian(s) if the patient is ≥ 9 to < 18 years old. An additional informed assent form must be signed by patient if ≥ 9 to <18 years old to confirm his willingness to participate in the study. If the patient becomes 18 years of age during the study, the patient must provide written informed consent at that time to continue study participation
2. Sex and age: Male and female patients aged ≥ 9 and <50 years
3. Diagnosis at screening and baseline visits:

   * a) Patients affected by facial acne vulgaris with: Investigator's Global Assessment (IGA) score:

     * equal to 3-4 if patient is > 14 and < 50 years old
     * ≥ 2 if the patient is ≥ 9 and ≤ 14 years old. Face Inflammatory lesions: ≥ 20 and ≤ 100 inflammatory lesions (papules and pustules) and ≤ 1 nodules on the face. Face Non-inflammatory lesions: ≥ 20 and ≤ 100 non-inflammatory lesions (open and closed comedones) on the face.
   * b) Patients affected also by truncal acne (optional criteria): The patient has a truncal acne on areas of the trunk (shoulders, upper back and upper anterior chest) accessible for patient's self-application of study medication with a severity grade equal to 2 or 3 on the Physician Global Assessment (PGA) scale. The patient has a minimum of 20 inflammatory lesions (papules and pustules) and 20 non-inflammatory lesions (open and closed comedones) but no more than 100 non-inflammatory lesions and no more than 100 inflammatory lesions and ≤ 1 nodules on areas of the trunk (shoulders, upper back and upper anterior chest) reachable to patient's self-application of study medication at screening and baseline
4. Full comprehension: Patients and their parents/legal guardian(s) (for <18 years old patients) can comprehend the whole nature and purpose of the study, including possible risks and side effects, and are able to cooperate with the Investigator and to comply with the requirements of the entire study
5. Contraception and fertility: Women of childbearing potential must be using an effective contraception method during the entire duration of the study (effective contraception methods are those considered at least "acceptable" according to CTFG Recommendations). A prior stable treatment period is required for the following reliable methods of contraception:

   * Hormonal oral, implantable, transdermal, or injectable contraceptives must be stable for at least 6 months before the baseline visit
   * A non-hormonal intrauterine device (IUD) must be started at least 2 months before the baseline visit.

Exclusion Criteria:

1. Acne:

   * Patients with a known history of acne persistent and unresponsive to topical and/or oral treatments within 6 months before randomization
   * Patients with generalized or localized acne forms other than acne vulgaris, e.g., acne conglobata, acne fulminans, acne rosacea, secondary acne (chloracne, drug-induced acne, etc), nodule-cystic acne
   * Patients with acne requiring systemic treatment
2. Beard and facial/body hair, tattoos:

   * Patients with a beard or who intend to grow a beard and/or to perform a facial tattoo during the study
   * Patients with facial hair or facial tattoos that could interfere with study assessments in the investigator's opinion
   * For patients with truncal acne: body hair, tattoos (or who intend to perform them) on the shoulders, upper back or upper anterior chest accessible to self-application of study medication by the patient (evaluable area) that may interfere with the study assessments in the investigator's opinion
3. Skin diseases: Patients with other active skin diseases (e.g., urticaria, atopic dermatitis, sunburn, seborrheic dermatitis, perioral dermatitis, rosacea, skin malignancies) or active skin infections in the facial or truncal region (bacterial, fungal, or viral) or any other facial or truncal disease or condition that might interfere with the evaluation of acne or place the patient at unacceptable risk
4. Allergy: Known or suspected hypersensitivity to any active or inactive ingredient in the study medications. Patients with a history of an allergic reaction or significant sensitivity to the formulations' ingredients
5. Topical therapies: Patients who are currently using, will use during the study, or discontinued less than 4 weeks before study baseline the use of prescribed and/or over-the-counter topical therapies for the treatment of acne, including but not limited to: corticosteroids, antibiotics, azelaic acid, benzoyl peroxide, salicylates, α-hydroxy/glycolic acid, any other topical cosmetic therapy for acne and retinoids on the face/trunk
6. Topical skin care products and procedures: Patients who are currently using, will use during the study, or discontinued less than 4 weeks before study baseline the use of products for facial/truncal application containing glycolic or other acids, masks, washes or soaps containing benzoyl peroxide or salicylic acid, non-mild cleansers or moisturizers containing retinol, salicylic or alpha- or beta-hydroxy acids, facial/truncal procedures such as chemical peel, laser treatment, photodynamic therapy, acne surgery, cryodestruction or chemodestruction, x-ray therapy, intralesional steroids, dermabrasion
7. Phototherapy: Patients who are currently using, will use during the study, or discontinued less than 4 weeks before study baseline phototherapy for the treatment of acne, including but not limited to: UV-A, UV-B, heliotherapy. Patients who have the need or plan to be exposed to artificial tanning devices or excessive sunlight during the study
8. Systemic therapies: Patients who are currently using, will use during the study, or discontinued less than 12 weeks before study baseline the use of systemic therapies for the treatment of acne, including but not limited to: antibiotics, isotretinoin. Other systemic therapies that could affect the patient's acne (i.e., anabolics, lithium, EGRF inhibitors, iodides, systemic corticosteroids - except inhaled corticosteroids or intrathecal corticosteroids - or other immunosuppressants), in the opinion of the investigator
9. Known systemic diseases that can lead to acneiform eruptions:

   1. Increased androgen production. 1) Adrenal origin: e.g., Cushing's disease, 21-hydroxylase deficiency; 2) Ovarian origin: e.g., polycystic ovarian syndrome, ovarian hyperthecosis
   2. Cryptococcosis disseminated
   3. Dimorphic fungal infections
   4. Behçet's disease
   5. Systemic lupus erythematosus (SLE)
10. Investigative studies: Participation in the evaluation of any investigational product or device within 24 weeks before study baseline
11. Diseases: Patients with underlying uncontrolled or unstable conditions (including but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal and auto-immune), which, in the Investigator's opinion, could significantly compromise the patient's safety and/or place the patient at an unacceptable risk. Any condition that in the investigator's opinion would make it unsafe for the patient to participate in the study.
12. Alcohol and other substance abuse: History of alcohol or other substance abuse within one year before screening
13. Communication: Patient(s) and parents/legal guardian(s) (if applicable) unable to communicate or cooperate with the investigator due to e.g., language problems, impaired cerebral function, impaired mental conditions
14. Reliability: Patients who may be unreliable for the study including patients who are unable to return for the scheduled visits
15. Pregnancy: Pregnant or breastfeeding women or women of childbearing potential who are planning to become pregnant during the study. *For all female patients of childbearing potential, pregnancy test result must be negative at screening.

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The relative change from baseline in total lesion count (inflammatory plus non-inflammatory) at V5/Wk12 on the face | From enrollment to the end of treatment at 12 weeks
Proportion of patients with an IGA success (face) at V5/Wk12. | From enrollment to the end of treatment at 12 weeks
  IGA success is defined according to the patient's age as:
  * a score of "clear" (score = 0) or "almost clear" (score = 1) for patients aged ≥ 9 and ≤ 14 years
  * a score of "clear" (score = 0) or "almost clear" (score = 1) in IGA at V5/Wk12 for patients aged > 14 and < 50 years.

SECONDARY OUTCOMES:
Absolute change from baseline in total lesion count at V5/Wk12 (face) | From enrollment to the end of treatment at 12 weeks
Percentage of patients who achieve an IGA success over the study duration (face) | From enrollment to the end of treatment at 12 weeks
  The Investigator Global Assessment (IGA) for acne is a 5-point clinical scale (0-4) used by dermatologists to assess overall acne severity based on lesion type and extent. It ranges from 0 (clear) to 4 (severe), providing a rapid, qualitative snapshot of facial acne, commonly used to measure treatment efficacy.
Change from baseline in total lesion count over the study duration (face) | From enrollment to the end of treatment at 12 weeks
Change from baseline in inflammatory lesion count over the study duration (face) | From enrollment to the end of treatment at 12 weeks
Change from baseline in non-inflammatory lesion count over the study duration (face) | From enrollment to the end of treatment at 12 weeks
Absolute change from baseline in total lesion count at V5/Wk12 (trunk) | From enrollment to the end of treatment at 12 weeks
Percentage of patients who achieve a PGA score of 1 (almost clear) or 0 (clear) and at least a two-grade improvement from baseline over the study duration | From enrollment to the end of treatment at 12 weeks
  The Physician Global Assessment (PGA) for acne is a standardized 5-point scale (0-4) used by clinicians to assess acne severity based on the number and type of lesions. It is frequently used in clinical trials and practice to measure treatment success, with a score of "clear" (0) or "almost clear" (1) usually indicating a successful outcome.
Change from baseline in truncal total lesion total count over the study duration | From enrollment to the end of treatment at 12 weeks
Change from baseline in truncal inflammatory lesion count over the study duration | From enrollment to the end of treatment at 12 weeks
Change from baseline in truncal non-inflammatory lesion count over the study duration. | From enrollment to the end of treatment at 12 weeks

OTHER OUTCOMES:
Dermatology Life Quality Index (DLQI) completed by the patient at the Baseline and Week 12/EoT visits | From enrollment to the end of treatment at 12 weeks
  The Dermatology Life Quality Index (DLQI) is a 10-question validated questionnaire used to measure the impact of skin diseases on a patient's life over the past week. Scores range from 0 to 30; higher scores indicate greater impairment.
Children's Dermatology Life Quality Index (C-DLQI for patients from 9 to 16 years old), completed by the patient at the Baseline and Week 12/EoT visits | From enrollment to the end of treatment at 12 weeks
  The Children's Dermatology Life Quality Index (CDLQI) is a 10-question validated questionnaire (ages 4-16) that measures skin disease impact on a child's life over the past week. Total scores range from 0-30, with higher scores indicating greater impairment
SCAR-S Scar Assessment at the Baseline and Week 12/EoT visits | From enrollment to the end of treatment at 12 weeks
  The Global Scale for Acne Scar Severity (SCAR-S) is a 6-point (0-5) clinician-reported system that grades acne scarring on the face, chest, and back. It classifies severity from 0 (clear) to 5 (very severe/prominent scarring) to evaluate the impact of atrophic or hypertrophic scars.
At selected sites: Photographic Scar Monitoring (not mandatory, following specific consent) at the Baseline and Week 12/EoT visits. | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (29):
- Italy (8):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona, AN
  - Azienda USL Toscana Centro, Florence, FI
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - Azienda Ospedaliero Universitaria Parma, Parma, PR
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Azienda Ospedaliera Policlinico Universitario Tor Vergata, Roma, RM
  - I.F.O. Istituti Fisioterapici Ospitalieri, Roma, RM
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, Napoli
- Poland (14):
  - Vitamed Galaj I Cichomski Sp. j., Bydgoszcz
  - DERMAPOLIS Medical Dermatology Center dr n.med. Edyta Gebska, Chorzów
  - Provita Sp. z o.o., Katowice
  - Silmedic Sp. z o.o., Katowice
  - Dermed Centrum Medyczne Sp. z o.o., Lodz
  - St-Inspire Sp. z o.o., Mikołów
  - Twoja Przychodnia Nowosolskie Centrum Medyczne Sp. z o.o., Nowa Sól
  - Labderm Essence Sp. z o.o., Ożarowice
  - Twoja Przychodnia Poznanskie Centrum Medyczne Sp. z o.o., Poznan
  - Lukmed 2 Sp. z o.o., Siedlce
  - Centrum Zdrowia Dziecka I Rodziny Im. Jana Pawla II W Sosnowcu Sp. z o.o., Sosnowiec
  - Klinika Ambroziak Sp. z o.o., Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - EMC Instytut Medyczny S.A., Wroclaw
- Spain (7):
  - Sant Joan De Deu Barcelona Hospital, Esplugues de Llobregat
  - Futuremeds Spain S.L., Madrid
  - Hospital Universitario Hm Sanchinarro, Madrid
  - Hospital Universitario Regional De Malaga, Málaga
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Quironsalud Infanta Luisa, Seville
  - Futuremeds Spain S.L., Seville